CLINICAL TRIAL: NCT00153075
Title: A Randomised Open Label, Six Way, Cross-over Scintigraphic Evaluation of the Effect of Inspiratory Flow Rate on Lung and Oropharyngeal Deposition With the Respimat Inhaler vs. a Metered Dose Inhaler (HFA-MDI) Using Berodual in Patients With Chronic Obstructive Pulmonary Disease (COPD).
Brief Title: Flow Rate Effect Respimat Inhaler Versus a Metered Dose Inhaler Using Berodual in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 215.1364
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Asthma
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma

INTERVENTIONS:
Device: Berodual Respimat
Device: Berodual HFA-MDI

SUMMARY:
The objective of this trial is to compare the total and regional deposition of aerosol in the lungs and oropharynx of patients with COPD at 3 different inspiratory flow rates following inhalation of Berodual delivered via the Respimat inhaler and Berodual? delivered via an HFA-metered dose inhaler.

DETAILED DESCRIPTION:
This is a single dose, randomised, active-controlled, six period, open-label cross-over trial in adult patients with COPD.

Berodual (fenoterol hydrobromide 50 g + ipratropium bromide 20 g) will be delivered via the Respimat inhaler and the MDI at 3 different inspiratory flow rates: 15 L/min, 30 L/min and 90 L/min. The optimal flow rate is expected to be 30 L/min for both inhalers.

On each test day patients will practise the inhalation manoeuvre with either a placebo Respimat or MDI inhaler. When patients can perform the inhalation technique correctly and they can obtain the required inspiratory flow rates the placebo will be replaced with the radio-labelled formulation.

The primary analysis will be carried out using the Sign Test. This is a non-parametric analysis in which no assumptions are made about the shape of the distribution of the responses from the Respimat inhaler and from the MDI under the null hypothesis.

Study Hypothesis:

The null hypothesis is that flow rate has the same effect on the Respimat and MDI inhalers. The alternative hypothesis is that flow rate has a different effect on the Respimat inhaler than on the MDI inhaler.

This means that under the null hypothesis the median of the differences between the Respimat inhaler and MDI pairs is zero i.e., the differences are equally lik ely to be positive or negative. Under the alternative hypothesis the median of the differences between the Respimat inhaler and MDI pairs is not zero i.e., the frequencies of the positive and negative signs are different.

Comparison(s):

For the primary comparison the whole lung deposition achieved for each patient at the 90 L/min flow rate will be expressed as a percentage of the whole lung deposition achieved by that patient at the 30 L/min flow rate for the Respimat and MDI inhalers separately. The difference between each pair of observations ((Respimat 90 L/min / Respimat 30 L/min) - (MDI 90 L/min / MDI 30 L/min)) will then be calculated and the sign of the direction of the difference noted i.e., positive or negative. The probability associated with the occurrence of the observed number of positive and negative differences will then be determined by reference to the binomial distribution with the probability of a positive or negative difference equal to 0.5 under the null hypothesis. If the alternative hypothesis is, however, true and flow rate does in fact have less effect on the Respimat inhaler than on the MDI inhaler, then there is likely to be a statistically significant greater number of positive differences.

ELIGIBILITY:
Inclusion Criteria:

* COPD patients:

  * FEV1 less or equal 65 % pre
  * FEV1 less or equal 70 % of FVC

Exclusion Criteria:

* Patients with any upper respiratory infection in the past 14 days prior to the Screening Visit (Visit 1)
* Patients with any unstable or life-threatening cardiac arrhythmia

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19
Dates: Start 2005-09-26 (Actual); Primary Completion 2005-12-07 (Actual); Study Completion 2005-12-07 (Actual)

PRIMARY OUTCOMES:
Whole lung deposition | 12 weeks

SECONDARY OUTCOMES:
Central lung zone deposition | 12 weeks
Intermediate lung zone deposition | 10 weeks
Peripheral lung zone deposition | 12 weeks
Ratio of peripheral to central zone deposition | 12 weeks
Oropharyngeal deposition | 12 weeks
Device deposition and exhaled air filter deposition | 12 weeks
FEV1 15, 30 and 60 minutes post-administration (safety only) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — B.I. Pharma GmbH & Co. KG
Locations (1):
- Inamed Research GmbH & Co. KG, Gauting, Germany